CLINICAL TRIAL: NCT00594425
Title: Photodynamic Therapy (PDT) With Methyl Aminolevulinate (MAL) Cream in Moderate to Severe Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PC TA202B/06
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — methyl 5-aminolevulinate; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): PDT using MAL concentration A
  Interventions: Drug: Methyl aminolevulinate (MAL) PDT
- 2 (Experimental): PDT using MAL concentration B
  Interventions: Drug: Methyl aminolevulinate (MAL) PDT
- 3 (Placebo Comparator): PDT using Placebo cream
  Interventions: Drug: Methyl aminolevulinate (MAL) PDT

INTERVENTIONS:
Drug: Methyl aminolevulinate (MAL) PDT — Cream application followed by illumination with red light

SUMMARY:
This multicenter study will be divided into 2 phases. The first phase will be an open label, dose-escalation phase, while the second will be a blinded, randomized, vehicle-controlled, parallel-group, dose-response phase. The second phase will only start if the first phase succeeds in establishing well tolerated dose(s). Patients with moderate to severe acne vulgaris in the face will be included.The results from part 2 has been presented in the result section.

DETAILED DESCRIPTION:
For the second part: All patients will receive 4 PDT sessions 2 weeks apart using a light dose of 37 J/cm2. One treatment group will receive vehicle cream, while the other 2 groups will receive MAL cream with a concentration of 40 mg/g and 80 mg/g, respectively. The MAL and vehicle cream will be applied in a thin layer on clean skin and left for 1.5 hours under occlusion before illumination.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients, age 15 to 40 years with moderate to severe facial acne vulgaris (IGA score 3-4).
2. Patients with skin type I to IV (Fitzpatrick).
3. Patients with 20 to 100 inflammatory lesions (papules, pustules, and nodules) on the face excluding lesions on the nose and in the peri-ocular area.
4. Patients with up to 200 noninflammatory lesions (open and closed comedones) on the face.
5. Patients with no more than 2 nodular lesions on the face.
6. Patients who are surgically sterile, postmenopausal, abstinent, or willing to use an adequate means of contraception including birth control pills, or barrier methods and spermicide for at least 14 days prior to Day 0. Patients using birth control pills must have used the same product and dose for at least 6 months and must agree to stay with the same product and dose for an additional 6 months.
7. Patients must be willing and capable of following study instructions to the extent and degree required by the protocol.
8. Patients must sign the approved informed consent form prior to any study procedures.
9. Patients must be willing to be photographed. Patients must be willing to sign a photography consent form.

Exclusion Criteria:

1. Known allergy to MAL, to a similar PDT compound, or to excipients of the cream.
2. Participation in other clinical studies either concurrently or within the last 30 days.
3. Patients who have a condition or who are in a situation, which, in the investigator's opinion, may put the patient at risk, may confound the study results, or may interfere with the patient's participation in the study.
4. Clinically significant sensitivity to visible light, or has porphyria or porphyrin sensitivity.
5. Exposure to ultraviolet radiation (UVB phototherapy, sun tanning salons) within the last 30 days.
6. Patients with a washout period for topical treatments for their acne of less than 14 days. Medicated cleansers may be used during the washout period and stopped before the treatment.
7. Patients with a washout period for oral antibiotics for treatment of their acne of less than 1 month.
8. Patients with a washout period for oral isotretinoin of less than 6 months.
9. Patients with a beard or other facial hair that might interfere with study assessments.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2007-02; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pariser, MD, Principal Investigator — AAD
Locations (14):
- United States (14):
  - Therapeutics Clinical Research, San Diego, California
  - Solano Clinical Research, Vallejo, California
  - DuPage Medical Group, Naperville, Illinois
  - Michigan Center for Research Corp, Clinton Twp, Michigan
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Associates of Rochester, Rochester, New York
  - Central Sooner Research, Norman, Oklahoma
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Dermatology Treatment & Research, Dallas, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - The Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient entered: February 07, 2007 Last patient last visit (12 week follow-up: July 07, 2008 Last patient last visit (24 week follow-up: September 22, 2008 15 medical derm clinics
Pre-assignment Details: Washout periods for prior acne treatment: 14 days for any topical treatment (except medicated cleansers), 1 month for oral antibiotics; 6 months for oral isotretinoin. Patients using birth control pills must have used the same product and dose for at least 6 months and had to agree to stay with the same product and dose for an additional 6 months.
Period: Overall Study
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Started | 50 | 48 | 52
Completed | 43 | 34 | 42
Not Completed | 7 | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT | Total
Number analyzed (Participants) | 50 | 48 | 52 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 17 | 11 | 39
  Between 18 and 65 years | 39 | 31 | 41 | 111
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 21.6 (5.24) | 20.2 (4.81) | 22.0 (5.00) | 21.3 (5.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 36 | 91
  Male | 22 | 21 | 16 | 59
Region of Enrollment [Number; unit: participants]
  United States | 50 | 48 | 52 | 150
Inflammatory lesion count [Mean (Full Range); unit: lesions] | 34.2 [20 to 81] | 32.1 [19 to 60] | 31.2 [20 to 74] | 32.5 [19 to 81]
Non inflammatory lesion count [Mean (Full Range); unit: lesions] | 39.1 [4 to 99] | 35.9 [5 to 111] | 35.2 [7 to 94] | 36.7 [4 to 111]
Investigator's Global Assessment (IGA) Score [Number; unit: participants]
  IGA SCORE 3 (MODERATE ACNE) | 35 | 41 | 44 | 120
  IGA SCORE 4 (SEVERE ACNE) | 15 | 7 | 8 | 30
Fitzpatrick Skin type [Number; unit: participants] — The patients is scored according to a predefined description of 4 different skin types.
  I White; very fair; red or blond hair; blue eyes; freckles Always burns, never tans
  II White; fair; red or blond hair; blue, hazel or green eyes Usually burns, tans with difficulty
  III Cream white; fair with any eye or hair color; very common Sometimes mild burn, gradually tans
  IV Brown; typical Mediterranean Caucasian skin Rarely burns, tans with ease
  participants
    Fitzpatrick skin type score I | 4 | 4 | 1 | 9
    Fitzpatrick skin type score II | 11 | 11 | 15 | 37
    Fitzpatrick skin type score III | 21 | 24 | 23 | 68
    Fitzpatrick skin type score IV | 14 | 9 | 13 | 36

OUTCOME MEASURES:

1. Secondary Outcome: Median Percentage Change in Facial Inflammatory (Nodules, Papules, and Pustules) Lesion Counts From Baseline
Time Frame: 3 weeks after last treatment
Population: PP population: excludes all patients with major protocol deviations (consists of the following types of events: Baseline inflammatory lesion count other than 20-100, received less that 4 treatments, primary efficacy criteria missing at week 12, insufficient primary efficacy follow up time, prohibited concomitant medication (retinoid).
Measure: Median (Full Range); unit: Percentage change
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 40 | 33 | 42
Percentage change | -44.5 (39,32) [-89 to 42] | -56.0 (44-34) [-95 to 44] | -40.5 (34-41) [-100 to 71]

2. Secondary Outcome: Median Percentage Change in Facial Inflammatory (Nodules, Papules, and Pustules) Lesion Counts From Baseline
Time Frame: 6 weeks after last treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: Percentage change
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 40 | 33 | 42
Percentage change | -52.0 [-92 to 88] | -69.5 [-95 to 45] | -52.0 [-96 to 71]

3. Secondary Outcome: Median Percentage Change in Facial Non Inflammatory Lesion Counts From Baseline
Time Frame: 6 weeks after last treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: Percentage change
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 40 | 33 | 42
Percentage change | -38.5 [-89 to 160] | -48.0 [-95 to 104] | -38.0 [-100 to 225]

4. Primary Outcome: Proportion of Success, Defined as Improvement of at Least 2 Grades From Baseline According to the IGA Scale Based on Facial Assessment
Time Frame: 12 weeks after last treatment
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 50 | 48 | 52
Percentage of participants | 16 [8.34 to 28.51] | 14.58 [7.25 to 27.17] | 11.54 [5.40 to 22.97]
Statistical Analysis 1: Comparison: 40 mg/g MAL PDT vs Vehicle PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.5288, Cochran-Mantel-Haenszel — Priori threshold for statistical significance was 5%; Cochran-Mantel-Haenszel test stratified by center. No adjustment for multiple comparisons was done; % success rate = 5.53, 95% CI 2-sided [-7.97 to 19.04]
Statistical Analysis 2: Comparison: 80 mg/g MAL PDT vs Vehicle PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.7539, Cochran-Mantel-Haenszel — Priori threshold for statistical significance was 5%; Cochran-Mantel-Haenszel test stratified by center. No adjustment for multiple comparisons was done; % success rate = 3.95, 95% CI 2-sided [-8.79 to 16.69]

5. Primary Outcome: Change in Facial Inflammatory (Nodules, Papules, and Pustules) Lesion Counts
Time Frame: 12 weeks after last treatment
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: lesions
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 50 | 48 | 52
lesions | -10.72 [-14.45 to -6.99] | -9.27 [-13.25 to -5.3] | -8.08 [-11.8 to -4.6]
Statistical Analysis 1: Comparison: 40 mg/g MAL PDT vs Vehicle PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.3236, ANCOVA — Priori threshold for statistical significance was 5%; ANCOVA model including center and baseline lesion count as a covariates. No adjustment for multiple comparisons was done; Least squares mean = -2.64, 95% CI 2-sided [-7.91 to 2.63]
Statistical Analysis 2: Comparison: 80 mg/g MAL PDT vs Vehicle PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.6657, ANCOVA — Priori threshold for statistical significance was 5%; [statistical method as in outcome 5, analysis 1]; Least squares mean = -1.19, 95% CI 2-sided [-6.64 to 4.26]

6. Secondary Outcome: Percent Reduction in Total Lesion Counts From Baseline
Time Frame: 6 weeks after last treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: Percentage change
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 38 | 32 | 41
Percentage change | -40 [-88 to 66] | -54 [-87 to 68] | -37 [-94 to 100]

7. Secondary Outcome: Proportion of Success, Defined as Improvement of at Least 2 Grades From Baseline According to the IGA Scale Based on Facial Assessment
Time Frame: 6 weeks after last treatment
Population: as for outcome 1
Measure: Number; unit: Precentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 42 | 40 | 33
Precentage of participants | 10.5 | 18.8 | 12.2

8. Secondary Outcome: The Proportion of Patients Rated as Clear or Almost Clear at 12 Weeks After Last Treatment
Time Frame: 12 weeks after last treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 40 | 33 | 42
percentage of participants | 10.0 | 18.2 | 11.9

9. Secondary Outcome: Facial Pain Using Visual Analouge Scale From 0 to 10, Were 0 Indicates no Pain and 10 Indicates Worst Pain.
Description: Measure was assessed on a Visual Analogue Scale from 0 to 10 cm
Time Frame: immediately after illumination-first treatment
Population: Safety
Measure: Median (Full Range); unit: cm
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 50 | 48 | 52
cm | 2.05 [0.0 to 10.0] | 2.25 [0.0 to 9.0] | 0.00 [0.0 to 3.5]

10. Secondary Outcome: Facial Pain Using Visual Analouge Scale From 0 to 10, Were 0 Indicates no Pain and 10 Indicates Worst Pain
Description: Measure was assessed on a Visual Analogue Scale from 0 to 10 cm
Time Frame: immediately after second treatment
Population: Safety
Measure: Mean (Full Range); unit: cm
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 46 | 41 | 50
cm | 2.0 [0.0 to 7.5] | 3.0 [0.0 to 8.0] | 0.0 [0.0 to 2.0]

11. Secondary Outcome: Facial Pain Using Visual Analouge Scale From 0 to 10, Were 0 Indicates no Pain and 10 Indicates Worst Pain.
Description: Measure was assessed on a Visual Analogue Scale from 0 to 10 cm
Time Frame: immediately after third treatment
Population: Safety
Measure: Median (Full Range); unit: cm
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 46 | 38 | 48
cm | 1.5 [0.0 to 8.0] | 2.0 [0.0 to 6.0] | 0.0 [0.0 to 1.0]

12. Secondary Outcome: Facial Pain Using Visual Analouge Scale From 0 to 10, Were 0 Indicates no Pain and 10 Indicates Worst Pain.
Description: Measure was assessed on a Visual Analogue Scale from 0 to 10 cm
Time Frame: immediately after illumination-fourth treatment treatment
Population: Safety
Measure: Median (Full Range); unit: cm
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 45 | 37 | 46
cm | 1.10 [0.0 to 6.4] | 2.50 [0.0 to 7.0] | 0.0 [0.0 to 2.4]

13. Secondary Outcome: Proportion of Patients With Mild and Moderate Erythema After First Treatment
Time Frame: immediately after first treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 50 | 48 | 52
percentage of participants | 75.1 | 61.7 | 17.6

14. Secondary Outcome: Proportion of Patients With Mild and Moderate Erythema After First Treatment
Time Frame: 2 days after first treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 50 | 48 | 52
percentage of participants | 44.9 | 44.7 | 17.6

15. Secondary Outcome: Proportion of Patients With Mild and Moderate Erythema After Second Treatment
Time Frame: immediately after second treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 50 | 48 | 52
percentage of participants | 67.4 | 65.8 | 18.0

16. Secondary Outcome: Proportion of Patients With Mild and Moderate Erythema After Third Treatment
Time Frame: immediately after third treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 50 | 48 | 52
percentage of participants | 67.4 | 71.1 | 16.7

17. Secondary Outcome: Proportion of Patients With Mild and Moderate Erythema After Fourth Treatment
Time Frame: immediately after fourth treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 50 | 48 | 54
percentage of participants | 45.9 | 63.1 | 15.2

18. Secondary Outcome: Proportion of Patients With Severe Erythema After First Treatment
Time Frame: immediately after first treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 50 | 48 | 52
percentage of participants | 0.0 | 2.1 | 0.0

19. Secondary Outcome: Proportion of Patients With Severe Erythema 2 Days After First Treatment
Time Frame: 2 days after first treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 49 | 47 | 51
percentage of participants | 2.0 | 0.0 | 0.0

20. Secondary Outcome: Proportion of Patients With Severe Erythema 7 Days After First Treatment
Time Frame: 7 days after first treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 50 | 46 | 51
percentage of participants | 2.0 | 0.0 | 0.0

21. Secondary Outcome: Proportion of Patients With Severe Erythema After Second Treatment
Time Frame: immediately after second treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 46 | 41 | 50
percentage of participants | 0.0 | 0.0 | 0.0

22. Secondary Outcome: Proportion of Patients With Severe Erythema After Third Treatment
Time Frame: immediately after third treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 46 | 38 | 48
percentage of participants | 0.0 | 0.0 | 0.0

23. Secondary Outcome: Proportion of Patients With Severe Erythema After Fourth Treatment
Time Frame: immediately after fourth treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 45 | 38 | 46
percentage of participants | 0.0 | 0.0 | 0.0

24. Secondary Outcome: Proportion of Patients With Mild and Moderate Hyperpigmentation After First Treatment
Time Frame: 2 days after treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 48 | 47 | 51
percentage of participants | 6.3 | 4.3 | 5.9

25. Secondary Outcome: Proportion of Patients With Mild and Moderate Hyperpigmentation After First Treatment
Time Frame: 2 weeks after first treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 49 | 46 | 51
percentage of participants | 2.0 | 10.8 | 5.9

26. Secondary Outcome: Proportion of Patients With Mild and Moderate Hyperpigmentation After Last Treatment
Time Frame: 2 weeks after last treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 46 | 38 | 45
percentage of participants | 8.6 | 21.1 | 4.4

27. Secondary Outcome: Proportion of Patients With Mild and Moderate Hyperpigmentation After Last Treatment
Time Frame: 6 weeks after last treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 44 | 37 | 43
percentage of participants | 6.8 | 8.1 | 9.3

28. Secondary Outcome: Proportion of Patients With Mild and Moderate Hyperpigmentation After Last Treatment
Time Frame: 12 weeks after last treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 45 | 38 | 45
percentage of participants | 4.4 | 5.3 | 6.7

29. Secondary Outcome: Proportion of Patients With Mild and Moderate Hypopigmentation After First Treatment
Time Frame: 2 days after first treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 48 | 47 | 51
percentage of participants | 2.1 | 0.0 | 0.0

30. Secondary Outcome: Proportion of Patients With Mild and Moderate Hypopigmentation After Last Treatment
Time Frame: 2 weeks after last treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 46 | 38 | 45
percentage of participants | 4.4 | 0.0 | 2.2

31. Secondary Outcome: Proportion of Patients With Mild and Moderate Hypopigmentation After First Treatment
Time Frame: 2 weeks after first treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 49 | 46 | 51
percentage of participants | 2.0 | 0.0 | 0.0

32. Secondary Outcome: Proportion of Patients With Mild and Moderate Hypopigmentation After Last Treatment
Time Frame: 6 weeks after last treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 44 | 37 | 43
percentage of participants | 2.3 | 2.7 | 0.0

33. Primary Outcome: Proportion of Success, Defined as Improvement of at Least 2 Grades From Baseline According to the IGA Scale Based on Facial Assessment
Time Frame: 12 weeks after last treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 42 | 40 | 33
percentage of participants | 17.5 [6.72 to 27.84] | 21.2 [8.75 to 31.95] | 16.7 [10.68 to 37.75]
Statistical Analysis 1: Comparison: 40 mg/g MAL PDT vs Vehicle PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.7889, Cochran-Mantel-Haenszel — Priori threshold for statistical significance was 5%; Cochran-Mantel-Haenszel stratified by center. No adjustment for multiple comparisons was done; %success rate = 3.09, 95% CI 2-sided [-11.16 to 17.33]
Statistical Analysis 2: Comparison: 80 mg/g MAL PDT vs Vehicle PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.8880, Cochran-Mantel-Haenszel — Priori threshold for statistical significance was 5%; Cochran-Mantel-Haenszel (CMH) test stratified by center. No adjustment for multiple comparisons was done; Percent success = 5.48, 95% CI 2-sided [-10.15 to 21.11]

34. Primary Outcome: Change in Facial Inflammatory (Nodules, Papules, and Pustules) Lesion Counts From Baseline
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: lesions
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 42 | 40 | 33
lesions | -10.95 [-15.18 to -6.72] | -11.8 [-16.65 to -6.95] | -10.62 [-15.12 to -6.12]
Statistical Analysis 1: Comparison: 40 mg/g MAL PDT vs Vehicle PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.9151, ANCOVA — Priori threshold for statistical significance was 5%; [statistical method as in outcome 5, analysis 1]; Least squares mean = -0.33, 95% CI 2-sided [-6.53 to 5.86]
Statistical Analysis 2: Comparison: 80 mg/g MAL PDT vs Vehicle PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.7233, ANCOVA — Priori threshold for statistical significance was 5%; [statistical method as in outcome 5, analysis 1]; Least squares mean = -1.18, 95% CI 2-sided [-7.81 to 5.45]

35. Secondary Outcome: Proportion of Patients With Mild and Moderate Hypopigmentation After Last Treatment
Time Frame: 12 weeks after last treatment
Population: Safety
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Number analyzed (Participants) | 45 | 38 | 45
percentage of participants | 2.2 | 0.0 | 0.0

ADVERSE EVENTS:
Arm/Group | 40 mg/g MAL PDT | 80 mg/g MAL PDT | Vehicle PDT
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/48 | 0/52
Other Adverse Events (participants affected / at risk) | 50/50 | 46/48 | 38/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg/g MAL PDT (N=50) | 80 mg/g MAL PDT (N=48) | Vehicle PDT (N=52)
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 1 | 0 | 0
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg/g MAL PDT (N=50) | 80 mg/g MAL PDT (N=48) | Vehicle PDT (N=52)
APPLICATION SITE DISCOLOURATION (Skin and subcutaneous tissue disorders) | 3 | 7 | 3
APPLICATION SITE DRYNESS (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
APPLICATION SITE ERYTHEMA (Skin and subcutaneous tissue disorders) | 40 | 35 | 17
APPLICATION SITE EXFOLIATION (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
APPLICATION SITE IRRITATION (Skin and subcutaneous tissue disorders) | 31 | 26 | 4
APPLICATION SITE PAIN (Skin and subcutaneous tissue disorders) | 32 | 31 | 5
APPLICATION SITE PARAESTHESIA (Skin and subcutaneous tissue disorders) | 3 | 9 | 4
APPLICATION SITE PRURITUS (Skin and subcutaneous tissue disorders) | 13 | 10 | 5
APPLICATION SITE SCAB (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
APPLICATION SITE WARMTH (Skin and subcutaneous tissue disorders) | 2 | 0 | 4
INFLUENZA (Infections and infestations) | 0 | 1 | 4
NASOPHARYNGITIS (Infections and infestations) | 3 | 1 | 1
SEASONAL ALLERGY (Immune system disorders) | 0 | 3 | 1
SINUSITIS (Infections and infestations) | 0 | 4 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 | 3 | 9
Headache (Nervous system disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data from the study are free for publication. However if publication of the results may endanger adequate patent protection for new principles,compounds,or formulations,Photocure has the right to decide when the results are free to be published. Before this agreed time, no data from the trial will be published, presented, or communicated, except to regulatory authorities and ethics committees. Both the investigators and Photocure will be given 30 days to review and comment.